CLINICAL TRIAL: NCT03766906
Title: STEM Familia Talk: A Bilingual Language Acquisition Smart Speaker App to Improve Academic Vocabulary, Engagement and Long-term Education and Health Outcomes for Latino Students and Their Families
Brief Title: STEM (Science, Technology, Engineering & Math) Familia Talk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MD013619-01; R44MD013619 (NIH)
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Language Development

STUDY DESIGN:
Intervention Model Description: One-arm, single-group, feasibility study with parent/student dyads.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Talk STEM Familia App (Experimental): This arm will test the feasibility of the Talk STEM Familia app to improve English language acquisition and family engagement and promote long-term educational and health outcomes among first- and second-generation Latino families.
  Interventions: Behavioral: Talk STEM Familia app

INTERVENTIONS:
Behavioral: Talk STEM Familia app — The Talk STEM Familia app will be used to improve access to sound instruction in scientific academic vocabulary through the development of a technology-enhanced, culturally responsive smart-speaker tool that engages Latino families in culturally responsive academic language acquisition and practice in the home setting.

SUMMARY:
After development of the Talk Stem Familia (TSF) smart-speaker application prototype, the study will evaluate the prototype's efficacy in a within-subjects pre-post design study. The sample will contain 50 parent-student/child dyads who will use the Alexa skill app for 6 weeks.

DETAILED DESCRIPTION:
Participants will receive an Echo Dot device enabled with the application prototype using a research Amazon account created for each dyad. The Echo Dot devices will be preconfigured by project staff onto research Amazon accounts. Parents will come to one of several orientation sessions to obtain their device and set-up instructions; staff will provide follow-up phone support as needed. Usage data will show how much the device is used by each dyad. To ensure exposure to TSF, parents will be asked to engage at least 3 times per week; project staff will prompt parents bi-weekly (via text, email, device notification, phone) during the 6-week intervention to encourage usage and provide needed technical support.

ELIGIBILITY:
Inclusion Criteria:

* Latino parents and their children who are students in grades 3 through 6.
* Parents have Spanish as primary home language.
* Family has wi-fi in the home.
* No age limits for parents. Their child must be in grades 3 through 6.

Exclusion Criteria:

* Parents and their children who are students in grade levels below grade 3 or above grade 6.
* Parents do not have Spanish as primary home language.
* Family does not have wi-fi in the home.
* Children younger than 8 (or in grade levels below grade 3).

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Smith, PhD, Study Chair — Oregon Research Behavioral Intervention Strategies, Inc.
Locations (1):
- Oregon Research Behavioral Intervention Strategies, Inc., Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Talk STEM Familia App
Started | 50 (50 dyads = 100 unique participants.)
Completed | 44 (44 dyads = 88 unique participants.)
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Population: Latinx, English-learner, parent/student dyads.
Arm/Group | Talk STEM Familia App
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants] — Parent participants reported age in years on demographic survey. Student participants had to be in 3rd -6th grade to be eligible to participate. Age was extrapolated from grade-level.
  Participants
    <=18 years | 50
    Between 18 and 65 years | 50
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline participants were 50 parent-student dyads, 50 parents and 50 students. Parent and student data were analyzed separately.
  Participants
    Student participants: number analyzed (Participants) | 50
    Student participants: Female | 29
    Student participants: Male | 21
    Parent participants: number analyzed (Participants) | 50
    Parent participants: Female | 44
    Parent participants: Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race/ethnicity information was only collected from parent participants.
  Participants
    Parent race/ethnicity: number analyzed (Participants) | 50
    Parent race/ethnicity: Euro American/Caucasian | 7
    Parent race/ethnicity: African American/Black | 2
    Parent race/ethnicity: American Indian or Alaskan Native | 1
    Parent race/ethnicity: More than one race | 28
    Parent race/ethnicity: Prefer not to disclose | 12

OUTCOME MEASURES:

1. Primary Outcome: Student Academic Vocabulary Knowledge in English
Description: The Student Academic Vocabulary Knowledge in English measure includes 18 multiple choice questions on the 18 words taught in the TSF app. The student chooses the correct word meaning from among four (4) possible responses. Students receive one point for each word correctly identified and points are summed across the 18 items. Scores can range from 0-18 and a higher score indicates greater vocabulary knowledge.
Time Frame: Baseline (pretest) and 6 weeks (posttest)
Population: Latinx, English-learner students.
Measure: Mean (Standard Deviation); unit: Number of correct responses
Arm/Group | Talk STEM Familia App
Number analyzed (Participants) | 50
Number of correct responses
  Pretest | 9.36 (3.71)
  Posttest | 11.39 (3.87)
Statistical Analysis 1: Comparison: Talk STEM Familia App; Test type: Superiority; p = .003, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = 2.03 — Investigators tested whether pretest to posttest change was significantly greater than 0 at P < 0.05

2. Primary Outcome: Parent Academic Vocabulary Knowledge in Spanish
Description: The Parent Academic Vocabulary Knowledge in Spanish measure includes 18 multiple choice questions on the 18 words taught in the TSF app. The parent chooses the correct word meaning from among four (4) possible responses. Parents receive one point for each word correctly identified and points are summed across the 18 items. Scores can range from 0-18 and a higher score indicates greater vocabulary knowledge.
Time Frame: Baseline (pretest) and 6 weeks (posttest)
Population: Latinx English learner parents
Measure: Mean (Standard Deviation); unit: Number of correct responses
Arm/Group | Talk STEM Familia App
Number analyzed (Participants) | 50
Number of correct responses
  Pretest | 12.40 (3.36)
  Posttest | 13.58 (3.11)
Statistical Analysis 1: Comparison: Talk STEM Familia App; Test type: Superiority; p = .022, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = 1.18 — Investigators tested whether pre-test to post-test change was significantly greater than zero at P<0.05

3. Primary Outcome: Student Academic Vocabulary Usage in English
Description: The Student Academic Vocabulary Usage in English measure includes 18 true/false questions testing student knowledge of correct usage of the 18 academic vocabulary words taught in the TSF app.
Time Frame: Baseline (pretest) and 6 weeks (posttest)
Population: Latinx, English-learner students.
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Talk STEM Familia App
Number analyzed (Participants) | 50
percentage of correct responses
  Pre-test | 12.14 (3.01)
  Post-test | 13.48 (2.95)
Statistical Analysis 1: Comparison: Talk STEM Familia App; Test type: Superiority; p = .016, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = 1.34 — Investigators tested whether pre-test to post-test change was significantly greater than 0 at P<0.05

4. Primary Outcome: Parent Academic Vocabulary Usage in Spanish
Description: The Parent Academic Vocabulary Usage in Spanish measure includes 18 true/false questions testing student knowledge of correct usage of the 18 academic vocabulary words taught in the TSF app.
Time Frame: Baseline (pretest) and 6 weeks (posttest)
Population: Latinx, English-learner parents.
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Talk STEM Familia App
Number analyzed (Participants) | 50
percentage of correct responses
  Pre-test | 14.08 (2.58)
  Post-test | 15.03 (1.96)
Statistical Analysis 1: Comparison: Talk STEM Familia App; Test type: Superiority; p = .002, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = 0.95 — Investigators tested whether pre-test to post-test change was significantly greater than 0 at P<0.05

5. Secondary Outcome: Student Engagement Instrument
Description: The Student Engagement Instrument (SEI; Betts, Appleton, Reschly, et al., 2010) consists of three subscales (future aspirations and goals, 5 items, r = .80, family support for learning, 6 items, r = .79, and control and relevance of school work, 9 items, r = 70). The SEI scale for each item ranges from 1-"Strongly disagree" to 5- "Strongly agree" with 5 indicating greater self-efficacy (more positive). A sum score was computed for each subscale. For future aspirations the scores can range from 5 to 25 and a higher score indicates a more positive outcome; greater self-efficacy for future aspirations. For family support for learning the score can range from 6 to 30 and a higher scores indicates a more positive outcome; greater self-efficacy for family support for learning. For control and relevance of school work the scores can range from 9 to 45 and a greater score indicates a more positive outcome; greater self-efficacy for control and relevance of school work.
Time Frame: Baseline (pretest) and 6 weeks (posttest)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Talk STEM Familia App
Number analyzed (Participants) | 50
score on a scale
  Relevance to schoolwork pre-test | 35.68 (5.93)
  Relevance to schoolwork post-test | 36.06 (5.17)
  Future aspirations pre-test | 21.78 (2.94)
  Future aspirations post-test | 21.73 (2.76)
  Family support pre-test | 25.18 (3.88)
  Family support post-test | 25.11 (3.66)
Statistical Analysis 1: Comparison: Talk STEM Familia App; The statistical analyses for the Student Self-Efficacy, in terms of type of statistical test, method, and the comments which we state within-subjects paired t-tests, are the same for each of the three subscales that make up Student Self-Efficacy (i.e., Relevance to schoolwork, Future aspirations, and Family support); Test type: Superiority; p = .626, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = 0.38 — Investigators tested whether pre-test to post-test change was significantly greater than 0 at P<0.05
Statistical Analysis 2: Comparison: Talk STEM Familia App; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = .909, t-test, 2 sided; Investigators tested whether pre-test to post-test change was significantly greater than 0 at P<0.05; Mean Difference (Final Values) = 0.05
Statistical Analysis 3: Comparison: Talk STEM Familia App; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = .905, t-test, 2 sided; Mean Difference (Final Values) = 0.07 — Investigators tested whether pre-test to post-test change was significantly greater than 0 at P<0.05

6. Secondary Outcome: The Efficacy to Influence School-related Performance Subscale of the Parental Self-Efficacy Scale
Description: The Efficacy to Influence School-related Performance subscale of the Parental Self-Efficacy Scale (PSES; Bandura, et al., 2001) (completed in Spanish) to measure useful factors that reflect parents' perceptions of whether they can influence their child's academic performance. The PSES consists of 8 items on a 9-point scale ranging from 1 = "nothing" to 9 = "a great deal" . The measure has an internal reliability of .87. A mean composite score was computed and the scores can range from 1 to 9 with a higher score indicating a more positive outcome; greater levels of self-efficacy.
Time Frame: Baseline (pretest) and 6 weeks (posttest)
Population: Latinx, English-learner parents.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Talk STEM Familia App
Number analyzed (Participants) | 50
score on a scale
  Parental Self-Efficacy at pre-test | 7.26 (1.19)
  Parental Self-Efficacy at post-test | 7.62 (1.08)
Statistical Analysis 1: Comparison: Talk STEM Familia App; Test type: Superiority; p = .054, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = 0.36 — Investigators tested whether pre-test to post-test change was significantly greater than 0 at P<0.05

7. Secondary Outcome: Student Academic Language Learning Behaviors
Description: The Student Academic Language Learning Behaviors measure includes 11 items asking students to estimate the frequency of discrete learning behaviors such as saying "scientific" words out loud in English and using "scientific" words in sentences. The measure uses a 4-point scale of frequency with 1 being "Not at all" and 4 being " 3-4 times a week." A sum score for the 11 items was computed and the scores could range from 11 to 44. Higher scores indicate a more positive outcome; greater frequency of behaviors.
Time Frame: Baseline (pretest) and 6 weeks (posttest)
Population: Latinx, English-learner students.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Talk STEM Familia App
Number analyzed (Participants) | 50
score on a scale
  Student academic language learning behavior at pre-test | 23.53 (7.65)
  Student academic language learning behavior at post-test | 27.01 (8.51)
Statistical Analysis 1: Comparison: Talk STEM Familia App; Test type: Superiority; p < .001, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = 3.48 — Investigators tested whether pre-test to post-test change was significantly greater than 0 at P<0.05

8. Secondary Outcome: Parent Academic Enabling Behaviors
Description: The Parent Academic Enabling Behaviors measure includes 13 items asking parents to estimate the frequency of their discrete academic enabling behaviors, such as helping their child learn the meaning of "scientific" words and using "scientific" words in a conversation with their child. The measure uses a 4-point scale of frequency with 1 being "Not at all" and 4 being " 3-4 times a week." A sum score including all 13 items was computed and can range between 13 and 52. Higher scores indicate a more positive outcome; greater frequency of behaviors.
Time Frame: Baseline (pretest) and 6 weeks (posttest)
Population: Latinx, English-learner students.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Talk STEM Familia App
Number analyzed (Participants) | 50
score on a scale
  Parent academic enabling behavior at pre-test | 18.24 (7.45)
  Parent academic enabling behavior at post-test | 25.76 (9.47)
Statistical Analysis 1: Comparison: Talk STEM Familia App; Test type: Superiority; p < .001, t-test, 2 sided; Within subjects paired t-tests; Mean Difference (Final Values) = 7.52 — Investigators tested whether pre-test to post-test change was significantly greater than 0 at P<0.05

ADVERSE EVENTS:
Description: No adverse events (Deaths, serious adverse events, and nonserious adverse events) were assessed or reported for study participants.
Arm/Group | Talk STEM Familia App
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT03766906/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT03766906/ICF_001.pdf